CLINICAL TRIAL: NCT03150277
Title: Post - Activation Potentiation Following Acute Bouts of Plyometric Versus Heavy Resistance Exercise in Collegiate Soccer Players
Brief Title: Post - Activation Potentiation After Plyometric and Heavy Resistance Exercise in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jamia Millia Islamia (Other)
Responsible Party: Principal Investigator, Md. Shahid Raza, Assistant Professor, Jamia Millia Islamia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 4/10/95/JMI/IEC/2016
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Soccer
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: Randomized crossover design
Who Masked: Participant
Masking Description: All the participants will be blinded about the knowledge of the outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric-Resistance (Experimental): This group will perform plyometric exercise first and then heavy resistance exercise
  Interventions: Behavioral: Plyometric exercise; Behavioral: Heavy resistance exercise
- Resistance-Plyometric (Experimental): This group will perform resistance exercise first and then plyometric exercise
  Interventions: Behavioral: Plyometric exercise; Behavioral: Heavy resistance exercise

INTERVENTIONS:
Behavioral: Plyometric exercise — 2 sets of 10 ankle hops, 3 sets of 5 hurdle hops, 5 drop-jumps from a height of 50 cm
Behavioral: Heavy resistance exercise — 10 single repetitions of back half squats at 90% of 1 repetition maximum

SUMMARY:
The main purpose of this study will be comparison of acute effects of plyometric and heavy resistance exercise on post-activation potentiation

DETAILED DESCRIPTION:
This is a single-center, randomized, crossover study. Collegiate soccer players will be enrolled in this study. The study will be performed in 3 separate sessions.In the first session, participants will be familiarized with the experimental conditions and 1RM will be calculated. Participants will then be randomized to receive either heavy resistance or plyometric exercise first in the second session and then will be crossed over to receive the opposite intervention in the third session. The objective of the study is to compare the acute effects of plyometric and heavy resistance exercise on post - activation potentiation by measuring physical performance and blood lactate level.

ELIGIBILITY:
Inclusion Criteria:

* Collegiate soccer players aged 18 - 26 years
* Participants must have at least 2 years of playing experience
* Participants should be involved in sport-specific training on at least 2 occasions per week and play competitively once per week

Exclusion Criteria:

* Lower extremity reconstructive surgery in last 24 months or unresolved musculoskeletal disorder which would prohibit subject to participate in the sport.
* Participants who are consuming (or had consumed) growth hormone, anabolic steroids or any kind of performance enhancing drugs.

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-05-13 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
Blood lactate level | Measured prior to and after the intervention period (at 1 minute and 10 minute)
  Small pinprick blood samples will be taken from fingertip and blood lactate level will be measured by Blood lactate analyser (EKF Diagnostic Lactate Scout +, UK). The area will be cleaned first, using a dry tissue to remove sweat, then an alcohol swab. Once the area is dry, the lancet (often with a spring loaded apparatus) will be used to pierce the skin.

SECONDARY OUTCOMES:
Countermovement jump height | Measured prior to and after the intervention period (at 1 minute and 10 minute)
  The countermovement jump height will be measured using an iPhone app 'My Jump'. Jump height will be determined using an acknowledged flight - time calculation. During the CMJ, the subject rest their hands on their hips while performing a downward movement, followed by a maximum effort vertical jump. The subjects have to land in an upright position and to bend knees on landing.
20 m single sprint time | Measured prior to and after the intervention period (at 1 minute and 10 minute)
  The 20m single sprint is a standard test for assessing soccer players' running speed. The test involves running a single maximum sprint over 20 meters, with the time recorded using a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Raza, MPT, Principal Investigator — Jamia Millia Islamia
Locations (1):
- Sports Complex, Jamia Millia Islamia, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No
Data will be kept secure with principal investigator (Md. Shahid Raza) and sub-investigator (Sourabh Kumar Sharma) due to confidentiality issues

REFERENCES:
- [Derived] Sharma SK, Raza S, Moiz JA, Verma S, Naqvi IH, Anwer S, Alghadir AH. Postactivation Potentiation Following Acute Bouts of Plyometric versus Heavy-Resistance Exercise in Collegiate Soccer Players. Biomed Res Int. 2018 Feb 7;2018:3719039. doi: 10.1155/2018/3719039. eCollection 2018. PMID 29568749